CLINICAL TRIAL: NCT05488236
Title: Embryo Ploidy Selection by Nuclear Magnetic Resonance: a Fast, Low Cost and Non-invasive Technique to Increase the Success Rate of ART
Brief Title: Nuclear Magnetic Resonance for Embryo Ploidy Selection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto Valenciano de Infertilidade de Lisboa (Network)
Collaborators: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Other Study IDs: 2004-LIS-037-SN
Record Dates: First submitted 2021-04-19; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Aneuploidy; Infertility
Keywords: Non-invasive embryo selection; Metabolic profile; Nuclear magnetic resonance
MeSH Terms: conditions — Aneuploidy; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples: culture medium from euploid and aneuploid embryos.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nuclear magnetic resonance analysis of embryo culture medium — Analysis of culture medium from euploid and aneuploid embryos by magnetic nuclear resonance.

SUMMARY:
This study aims to validate the embryo culture medium analysis by nuclear magnetic resonance spectroscopy, as a faster and less-costly alternative to preimplantation genetic test for aneuploidy which could significantly enhance embryo selection and the success rate of assisted reproductive technologies.

DETAILED DESCRIPTION:
Assisted reproductive technologies (ART) refers to treatments used to assist people in achieving a pregnancy. Over the last years, ART have been developed with efforts to deliver a healthy baby. However, the selection of the embryo that most likely results in pregnancy remains a critical step in ART. Currently, this selection is based on morphological assessment of the embryos, but up to 70% of those embryos display an abnormal number of chromosomes. Preimplantation genetic test for aneuploidy (PGT-A) is used to assess the ploidy of embryos, although this is an invasive, expensive and time consuming technique. Alternatively, in order to predict the ploidy of pre-implantation embryos (euploidy vs aneuploidy), we suggest to characterise the metabolic profile of the embryo culture medium by Nuclear Magnetic Resonance (NMR), which is a non-invasive, low cost and fast technique.

The aim of this study is to assess whether, using multivariable analysis to all the collected NMR data, it is possible to identify a differential metabolic pattern between aneuploid and euploid embryos which could improve embryo selection.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 and <49 years old.
* Body Mass Index ≥18.5 Kg/m2 and <30 Kg/m2.
* Planned for in vitro fertilization followed by preimplantation genetic test for aneuploidy.
* Oocytes retrieval and fertilization by intracytoplasmic sperm injection
* Six follicles over 14 mm on the day of the triggering. Gonadotropin-releasing hormone antagonist
* Signed and dated informed consent.

Exclusion Criteria:

* Previous history of poor ovarian response (<4 oocytes retrieved) with a maximal dose of ovarian stimulation (≥300 IU/day).
* Presence of a medical condition which is known to affect assisted reproductive technologies outcome (e.g. thyroid dysfunction).
* Active female smoking.
* Current use of anti-depressants, anti-psychotics, steroids, antiepileptics or chemotherapy.
* Those unable to comprehend the investigational nature of the proposed study.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Healthy women who will undergo a In vitro fertilization followed by preimplantation genetic test for aneuploidy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-10-07 (Estimated); Study Completion 2023-12-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the metabolites present in the culture medium of euploid versus aneuploid embryos. | 6 months
  The metabolites present in the culture medium of euploid and aneuploid embryos will be identified by NMR and compared to the metabolites present in the culture medium without embryo (control). The metabolic profiles of cultures form euploid and aneuploid embryos will be compared to the metabolic profile of culture medium without embryo.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Nunes, PhD, Principal Investigator — Instituto Valenciano de Infertilidade de Lisboa
Locations (1):
- Instituto Valenciano de Infertilidade, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No